CLINICAL TRIAL: NCT07140913
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of Adjunctive KarXT for the Treatment of Mania, With or Without Mixed Features, in Individuals With Bipolar-I Disorder Taking Lithium, Valproate, or Lamotrigine
Brief Title: A Study to Evaluate the Efficacy and Safety of Adjunctive KarXT for the Treatment of Mania, With or Without Mixed Features, in Participants With Bipolar-I Disorder Taking Lithium, Valproate, or Lamotrigine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0046; 2025-521845-26 (Other: EU CTR); U1111-1321-1513 (Other: WHO)
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mania; Bipolar Disorder
Keywords: Bipolar-I Disorder; Mania; KarXT; adjunctive treatment; mood stabilizer
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — xanomeline; trospium chloride; Lithium; Valproic Acid; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + Lithium, Valproate, or Lamotrigine (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Lithium; Drug: Valproate; Drug: Lamotrigine
- Placebo + Lithium, Valproate, or Lamotrigine (Placebo Comparator)
  Interventions: Drug: Lithium; Drug: Valproate; Drug: Lamotrigine; Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline/Trospium Chloride — Specified dose on specified days
  Other Names: KarXT; BMS-986510
  Arms: KarXT + Lithium, Valproate, or Lamotrigine
Drug: Lithium — Specified dose on specified days
Drug: Valproate — Specified dose on specified days
Drug: Lamotrigine — Specified dose on specified days
Drug: Placebo — Specified dose on specified days
  Arms: Placebo + Lithium, Valproate, or Lamotrigine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adjunctive KarXT for the treatment of mania in participants with Bipolar-I Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Individuals have a primary diagnosis of Bipolar-I disorder established by a comprehensive psychiatric evaluation based on the DSM-5-TR criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) version 7.0.2 Standard.
* Individual is experiencing an acute exacerbation or relapse of manic episode, with or without mixed features (≤ 3 weeks).
* The individual requires hospitalization for the acute exacerbation or relapse of mania.
* Body mass index ≥ 18 and ≤ 40 kg/m2
* Currently experiencing an acute episode of mania or mania with mixed features with a therapeutic dose of lithium, valproate, or lamotrigine. The dose of the mood stabilizer must have remained stable for at least two weeks prior to screening. Additionally, participants on valproate must have been receiving treatment with valproate for a minimum of seven months.
* YMRS Total Score of ≥ 18 at Screening and at Baseline, and < 20% reduction in YMRS from screening to baseline.
* Clinical Global Impression Severity scale (CGI-BP) ≥ 4

Exclusion Criteria:

* Any primary DSM-5-TR disorder other than BP-I within 12 months before screening (confirmed using MINI version 7.0.2 Standard) including BP-I depression, BP-I with rapid cycling, first manic episode, BP-II, and major depressive disorder.
* Individual has a DSM-5-TR diagnosis of moderate to severe substance use disorder (except tobacco use disorder) within the 12 months before screening (confirmed using MINI version 7.0.2 Standard at screening), or current use as determined by urine toxicology screen or alcohol test.
* Risk for suicidal behavior at screening as determined by the investigator's clinical assessment and the C-SSRS with an answer "Yes" to item 4 or 5 within 6 months before screening or between screening and baseline, or suicide attempt within 12 months before screening, or between screening and baseline
* History of irritable bowel syndrome (with or without constipation) or any serious constipation requiring treatment within the last 6 months.
* History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma.
* Participants with HIV, cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or the LFT results.
* Elevations in hepatic transaminases at screening ≥ 2 × ULN for ALT and AST and/or bilirubin > 1.5× ULN, unless in the context of Gilbert's syndrome.
* All grades of hepatic impairment (mild [Child-Pugh Class A], moderate [Child-Pugh Class B], and severe [Child-Pugh Class C]).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Young Mania Rating Scale (YMRS) at Week 5 | At Week 5

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impressions Bipolar (CGI-BP) at Week 5 | At Week 5
Occurrence of response at Week 5 assessed as the number of participants with a ≥ 50% decrease from baseline in Young Mania Rating Scale (YMRS) score | At Week 5
Occurrence of response at Week 5 assessed as the number of participants with a ≥ 1 change from baseline in CGI-BP | At Week 5
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 7
Number of participants with Serious Adverse Events (SAEs) | Up to Week 7
Number of participants with TEAEs leading to treatment discontinuation | Up to Week 5
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 7
Change from baseline in Barnes Akathisia Rating Scale (BARS) at Week 5 | At Week 5
Change from baseline in Simpson Angus Scale (SAS) at Week 5 | At Week 5
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) at Week 5 | At Week 5
Change from baseline in International Prostate Symptom Score (IPSS) at Week 5 | At Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (101):
- United States (20):
  - Pillar Clinical Research - Bentonville, Bentonville, Arkansas
  - Pillar Clinical Research- Little Rock, Little Rock, Arkansas
  - Clinical Innovations, Inc. dba CITrials, Bellflower, California
  - Inland Psychiatric Medical Group - Chino, Chino, California
  - Proscience Research Group, Culver City, California
  - Omega Clinical Trials - La Habra, La Habra, California
  - Catalina Research Institute, LLC, Montclair, California
  - NRC Research Institute, Orange, California
  - Clinical Innovations, Inc. dba CITrials, Riverside, California
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Health Synergy Clinical Research, Stuart, Florida
  - CenExel iResearch, LLC, Savannah, Georgia
  - Pillar Clinical Research -Chicago, Chicago, Illinois
  - Arch Clinical Trials, St Louis, Missouri
  - Richmond Behavioral Associates, Staten Island, New York
  - Community Clinical Research, Austin, Texas
  - Local Institution - 0160, Houston, Texas
  - Prime Clinical Research - Mansfield, Mansfield, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
- Argentina (6):
  - Local Institution - 0011, ABB, Buenos Aires F.D.
  - Local Institution - 0010, Córdoba
  - Local Institution - 0012, Córdoba
  - Local Institution - 0008, Córdoba
  - Local Institution - 0009, Mendoza
  - Local Institution - 0114, Santiago del Estero
- Bulgaria (6):
  - Local Institution - 0184, Kazanlak, Stara Zagora
  - Local Institution - 0124, Novi Iskar
  - Local Institution - 0084, Pleven
  - Local Institution - 0125, Plovdiv
  - Local Institution - 0181, Sliven
  - Local Institution - 0086, Targovishte
- China (11):
  - Local Institution - 0190, Beijing, Beijing Municipality
  - Local Institution - 0191, Guangzhou, Guangdong
  - Local Institution - 0193, Baoding, Hebei
  - Local Institution - 0187, Shijiazhuang, Hebei
  - Local Institution - 0196, Nanjing, Jiangsu
  - Local Institution - 0186, Xian, Shanxi
  - Local Institution - 0192, Chengdu, Sichuan
  - Local Institution - 0188, Tianjin, Tianjin Municipality
  - Local Institution - 0197, Ningbo, Zhejiang
  - Local Institution - 0185, Beijing
  - Local Institution - 0195, Changsha
- Denmark (3):
  - Local Institution - 0088, Hillerød, Capital Region
  - Local Institution - 0054, Aalborg, North Denmark
  - Local Institution - 0091, Glostrup Municipality
- France (5):
  - Local Institution - 0126, Nice, Alpes-Maritimes
  - Local Institution - 0085, Clermont-Ferrand, Puy-de-Dôme
  - Local Institution - 0087, Marseille
  - Local Institution - 0129, Montpellier
  - Local Institution - 0089, Paris
- India (4):
  - Local Institution - 0121, Mangalore, Karnataka
  - Local Institution - 0123, Madurai, Tamil Nadu
  - Local Institution - 0118, Kolkata, West Bengal
  - Local Institution - 0116, Kolkata
- Israel (5):
  - Local Institution - 0052, Hod HaSharon, Central District
  - Local Institution - 0050, Ramat Gan, Central District
  - Local Institution - 0053, Ashkelon, Southern District
  - Local Institution - 0199, Beersheba, Southern District
  - Local Institution - 0083, Jerusalem
- Italy (5):
  - Local Institution - 0003, Milan, Lombardy
  - Local Institution - 0005, Pisa, Tuscany
  - Local Institution - 0001, Siena, Tuscany
  - Local Institution - 0004, Ancona
  - Local Institution - 0002, Genova
- Japan (12):
  - Local Institution - 0173, Toyoake, Aichi-ken
  - Local Institution - 0172, Iizuka, Fukuoka
  - Local Institution - 0141, Kitakyushu-shi, Fukuoka
  - Local Institution - 0108, Sapporo, Hokkaido
  - Local Institution - 0107, Yokohama, Kanagawa
  - Local Institution - 0142, Kochi, Kochi
  - Local Institution - 0175, Karatsu, Saga-ken
  - Local Institution - 0180, Bunkyo-ku, Tokyo
  - Local Institution - 0139, Bunkyo-ku, Tokyo
  - Local Institution - 0201, Kodaira, Tokyo
  - Local Institution - 0176, tabashi City, Tokyo
  - Local Institution - 0174, Fukuoka
- Poland (2):
  - Local Institution - 0103, Rybnik, Silesian Voivodeship
  - Local Institution - 0082, Tuszyn, Łódź Voivodeship
- Romania (10):
  - Local Institution - 0102, Bucharest, București
  - Local Institution - 0092, Bucharest, București
  - Local Institution - 0093, Bucharest, București
  - Local Institution - 0094, Bucharest, București
  - Local Institution - 0098, Bucharest, București
  - Local Institution - 0096, Bucharest
  - Local Institution - 0099, Bucharest
  - Local Institution - 0097, Iași
  - Local Institution - 0095, Sanpetru /Brasov
  - Local Institution - 0101, Sibiu
- Ukraine (12):
  - Local Institution - 0167, Smila, Cherkasy Oblast
  - Local Institution - 0178, Skarzhyntsi, Khmelnytskyi Oblast
  - Local Institution - 0169, Hlevakha, Kyiv Oblast
  - Local Institution - 0162, Kyiv, Kyivska Oblast
  - Local Institution - 0164, Lviv, Lviv Oblast
  - Local Institution - 0177, Poltava, Poltava Oblast
  - Local Institution - 0168, Vinnytsia, Vinnytsia Oblast
  - Local Institution - 0165, Dnipropetrovsk
  - Local Institution - 0163, Kropyvnytskyi
  - Local Institution - 0170, Odesa
  - Local Institution - 0171, Odesa
  - Local Institution - 0166, Ternopil

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07140913.html